CLINICAL TRIAL: NCT03470376
Title: Lipid-lowering and Vascular Effects of a Nutraceutical Combination in HIV-infected Patients on Stable Antiretroviral Therapy
Brief Title: NUtraceutical TReatment for hYpercholesterolemia in HIV-infected Patients
Acronym: NU-TRY(HIV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Matteo Pirro, Clinical Professor, Principal Investigator, University Of Perugia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-006
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Hypercholesterolemia; Inflammation; Atherosclerosis
Keywords: cholesterol; nutraceutical; HIV; PCSK9; hsCRP; stiffness
MeSH Terms: conditions — Hypercholesterolemia; Inflammation; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: NC vs noNC
Who Masked: Outcomes Assessor
Masking Description: Patients names and allocation to arms was masked for outcomes assessors
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutraceutical combination (NC) (Experimental): Patients on standardized diet regimen taking a NC (red yeast rice-derived monacolin K 3 mg, berberine 500 mg, policosanol 10 mg, astaxanthin 0.5 mg, folic acid 0.2 mg and coenzyme Q10 2 mg) one pill/day for 3 months
  Interventions: Dietary Supplement: Nutraceutical combination (NC)
- No nutraceutical combination (noNC) (Active Comparator): Patients on standardized diet regimen without taking any NC
  Interventions: Behavioral: No nutraceutical combination (noNC)

INTERVENTIONS:
Dietary Supplement: Nutraceutical combination (NC) — An oral NC (red yeast rice-derived monacolin K 3 mg, berberine 500 mg, policosanol 10 mg, astaxanthin 0.5 mg, folic acid 0.2 mg and coenzyme Q10 2 mg) one pill/day was administered for 3 months along with prosecution of standardized diet regimen
  Other Names: Armolipid Plus, Meda Pharma - Mylan
  Arms: Nutraceutical combination (NC)
Behavioral: No nutraceutical combination (noNC) — Prosecution of standardized diet regimen for 3 months
  Arms: No nutraceutical combination (noNC)

SUMMARY:
The effects of a nutraceutical combination (NC) containing low-dose monacolin K and berberine on lipid profile, proprotein convertase subtilisin/kexin type 9 (PCSK9), subclinical inflammation and arterial stiffness were investigated in human immunodeficiency virus (HIV)-infected patients receiving stable antiretroviral therapy (ART).

DETAILED DESCRIPTION:
This is a crossover interventional study of 26 HIV-infected patients on stable ART with low density lipoprotein cholesterol (LDL-C) >100 mg/dL, not receiving any lipid-lowering treatment. After a 3-week lipid stabilization period with a standardized diet regimen, the effect of a 3-month oral NC containing red yeast rice-derived monacolin K 3 mg, berberine 500 mg, policosanol 10 mg, astaxanthin 0.5 mg, folic acid 0.2 mg and coenzyme Q10 2 mg vs no active treatment (noNC) was tested on plasma total cholesterol (TC), LDL-C, high density lipoprotein cholesterol (HDL-C), triglyceride, lipoprotein(a), PCSK9, high-sensitivity C-reactive protein (hsCRP) levels and aortic pulse wave velocity (aPWV).

ELIGIBILITY:
Inclusion Criteria:

* LDL-C >100 mg/dL
* no history of cardiovascular disease
* stable ART for at least 6 months

Exclusion Criteria:

* current or recent (≤6 months) treatment with lipid-lowering drugs
* chronic kidney disease [estimated glomerular filtration rate (GFR) <60 ml/min]
* liver impairment (AST and/or ALT >3 times upper limit of normal)
* current pregnancy
* opportunistic infections within the past 3 months,
* having received an organ transplant/immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL-C levels at 3 months | 3 months after treatment randomization
  plasma LDL-C levels

SECONDARY OUTCOMES:
Change from baseline in PCSK9 levels at 3 months | 3 months after treatment randomization
  plasma PCSK9 levels
Change from baseline in subclinical inflammation at 3 months | 3 months after treatment randomization
  plasma hs-CRP levels
Change from baseline in arterial stiffness at 3 months | 3 months after treatment randomization
  aPWV

OTHER OUTCOMES:
Change from baseline in creatine phosphokinase (CPK) levels at 3 months | 3 months after treatment randomization
  plasma CPK levels
Change from baseline in aspartate transaminase (AST) levels at 3 months | 3 months after treatment randomization
  plasma AST levels
Change from baseline in alanine transaminase (ALT) levels at 3 months | 3 months after treatment randomization
  plasma ALT levels
Change from baseline in CD4+ cell count at 3 months | 3 months after treatment randomization
  CD4+ cell count
Change from baseline in HIV-1 RNA levels at 3 months | 3 months after treatment randomization
  HIV-1 RNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Pirro, M.D., PhD, Principal Investigator — University Of Perugia

REFERENCES:
- [Background] Kelesidis T, Currier JS. Dyslipidemia and cardiovascular risk in human immunodeficiency virus infection. Endocrinol Metab Clin North Am. 2014 Sep;43(3):665-84. doi: 10.1016/j.ecl.2014.06.003. PMID 25169560
- [Background] Chastain DB, Stover KR, Riche DM. Evidence-based review of statin use in patients with HIV on antiretroviral therapy. J Clin Transl Endocrinol. 2017 Feb 22;8:6-14. doi: 10.1016/j.jcte.2017.01.004. eCollection 2017 Jun. PMID 29067253
- [Background] Bednasz C, Luque AE, Zingman BS, Fischl MA, Gripshover BM, Venuto CS, Gu J, Feng Z, DiFrancesco R, Morse GD, Ma Q. Lipid-Lowering Therapy in HIV-Infected Patients: Relationship with Antiretroviral Agents and Impact of Substance-Related Disorders. Curr Vasc Pharmacol. 2016;14(3):280-7. doi: 10.2174/1570161114666160106151652. PMID 26733388
- [Background] Pirro M, Vetrani C, Bianchi C, Mannarino MR, Bernini F, Rivellese AA. Joint position statement on "Nutraceuticals for the treatment of hypercholesterolemia" of the Italian Society of Diabetology (SID) and of the Italian Society for the Study of Arteriosclerosis (SISA). Nutr Metab Cardiovasc Dis. 2017 Jan;27(1):2-17. doi: 10.1016/j.numecd.2016.11.122. Epub 2016 Nov 22. PMID 27956024
- [Background] Pirro M, Mannarino MR, Ministrini S, Fallarino F, Lupattelli G, Bianconi V, Bagaglia F, Mannarino E. Effects of a nutraceutical combination on lipids, inflammation and endothelial integrity in patients with subclinical inflammation: a randomized clinical trial. Sci Rep. 2016 Mar 23;6:23587. doi: 10.1038/srep23587. PMID 27004462
- [Background] Barrios V, Escobar C, Cicero AF, Burke D, Fasching P, Banach M, Bruckert E. A nutraceutical approach (Armolipid Plus) to reduce total and LDL cholesterol in individuals with mild to moderate dyslipidemia: Review of the clinical evidence. Atheroscler Suppl. 2017 Feb;24:1-15. doi: 10.1016/j.atherosclerosissup.2016.10.003. Epub 2016 Dec 18. PMID 27998714
- [Background] Pirro M, Mannarino MR, Bianconi V, Simental-Mendia LE, Bagaglia F, Mannarino E, Sahebkar A. The effects of a nutraceutical combination on plasma lipids and glucose: A systematic review and meta-analysis of randomized controlled trials. Pharmacol Res. 2016 Aug;110:76-88. doi: 10.1016/j.phrs.2016.04.021. Epub 2016 May 6. PMID 27157250
- [Background] Keithley JK, Swanson B, Sha BE, Zeller JM, Kessler HA, Smith KY. A pilot study of the safety and efficacy of cholestin in treating HIV-related dyslipidemia. Nutrition. 2002 Feb;18(2):201-4. doi: 10.1016/s0899-9007(01)00688-8. PMID 11844656
- [Background] Kinlay S. Low-density lipoprotein-dependent and -independent effects of cholesterol-lowering therapies on C-reactive protein: a meta-analysis. J Am Coll Cardiol. 2007 May 22;49(20):2003-9. doi: 10.1016/j.jacc.2007.01.083. Epub 2007 May 4. PMID 17512355
- [Derived] Pirro M, Francisci D, Bianconi V, Schiaroli E, Mannarino MR, Barsotti F, Spinozzi A, Bagaglia F, Sahebkar A, Baldelli F. NUtraceutical TReatment for hYpercholesterolemia in HIV-infected patients: The NU-TRY(HIV) randomized cross-over trial. Atherosclerosis. 2019 Jan;280:51-57. doi: 10.1016/j.atherosclerosis.2018.11.026. Epub 2018 Nov 14. PMID 30471555